CLINICAL TRIAL: NCT05370885
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of VE202 in Patients With Mild-to-Moderate Ulcerative Colitis
Brief Title: VE202 in Patients With Mild-to-Moderate Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following review of Part 1 study data, the Sponsor decided to terminate the study with immediate effect. Results indicated that VE202 was not superior to placebo on the primary or any of the secondary endpoints. No new safety concerns were observed.
Sponsor: Vedanta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VE202-002; 2021-001280-24 (EudraCT Number)
Record Dates: First submitted 2022-03-30; First posted 2022-05-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis; Colitis, Ulcerative
Keywords: Ulcerative Colitis; VE202; Vedanta; Clostridia
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: Part 1 Active and Part 2 Placebo Treatment with Vancomycin pretreatment. (Other): In Part 1 of the study, patients in Group A will receive VE202 for 8 weeks.
  In Part 2 of the study, patients in Group A will receive VE202 placebo for 2 weeks.
  In Part 3, patients will be followed for safety for 1 year from the start of treatment.
  Interventions: Biological: VE202; Drug: Vancomycin Oral Capsule; Other: VE202 Placebo; Other: Vancomycin Placebo
- Group B: Part 1 Placebo and Part 2 Active Treatment with Vancomycin pretreatment. (Other): In Part 1 of the study, patients in Group B will receive VE202 placebo for 8 weeks.
  In Part 2 of the study, patients in Group B will receive VE202 for 2 weeks.
  In Part 3, patients will be followed for safety for 1 year from the start of treatment.
  Interventions: Biological: VE202; Drug: Vancomycin Oral Capsule; Other: VE202 Placebo; Other: Vancomycin Placebo

INTERVENTIONS:
Biological: VE202 — VE202 is a rationally defined, live biotherapeutic product for oral administration.
Drug: Vancomycin Oral Capsule — Vancomycin is an antibiotic used to treat or prevent infection
Other: VE202 Placebo — VE202 Placebo
Other: Vancomycin Placebo — Vancomycin Placebo

SUMMARY:
A Phase 2 study to evaluate the safety, efficacy, and microbiota changes of VE202 in patients with mild to moderate ulcerative colitis (UC).

DETAILED DESCRIPTION:
A Phase 2 double-blind, placebo-controlled, randomized study to evaluate the safety, efficacy, and microbiota changes of VE202 in biologic-naïve patients with mild to moderate UC. In Parts 1 and 2 of the study, patients will receive VE202 or placebo for 8 weeks or 2 weeks. In Part 3, patients will be followed for safety for 1 year from the start of treatment.

ELIGIBILITY:
KEY INCLUSION CRITERIA

1. 18 to 75 years of age
2. Documented clinical and endoscopic diagnosis of UC at least 3 months prior to randomization
3. Active mild to moderate UC, as defined by the following:

   1. Disease that extends at least 15 cm from the anal verge
   2. A modified Mayo score of 4 to 8 with: (i.) Mayo endoscopic subscore of ≥ 2 based on screening flexible sigmoidoscopy; (ii.) Rectal bleeding score of ≥ 1
4. Has never received a biologic agent, Janus kinase inhibitor, or sphingosine-1-phosphate modulator for the treatment of UC
5. If receiving corticosteroids, dose must be stable for at least 4 weeks before randomization
6. Doses of other allowable UC medications must be stable for at least 8 weeks before randomization

KEY EXCLUSION CRITERIA

1. Known history of Crohn's disease (CD) or indeterminate colitis
2. A known diagnosis of primary sclerosing cholangitis
3. Allergy to VE202 or any of its components
4. Allergy to vancomycin or any of its components
5. A diagnosis of any non-IBD diarrheal illness (eg, Clostridioides difficile, celiac disease, parasitic infection) within 3 months prior to randomization
6. Use of probiotics or herbal, botanical, or traditional medicinal preparations within the 2 weeks prior to randomization (consumption of food products such as yogurt, kefir, kombucha, and herbal teas is permissible)
7. Receipt of Fecal Microbiota Transplantation (FMT) or other fecal-derived preparation within 6 months prior to randomization
8. Prior colectomy, ostomy, or other intestinal surgery (excluding cholecystectomy or appendectomy)
9. Receipt of any investigational biologic within 60 days or 5 half-lives prior to randomization, whichever is longer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with endoscopic response on flexible sigmoidoscopy after 8 weeks of treatment with VE202 or placebo. | 8 Weeks
  Endoscopic response is defined as a reduction from baseline of 1 point or more in Mayo endoscopic subscore. The Mayo endoscopic subscore is evaluated on a scale of 0 to 3, with a higher score representing more severe disease.
Percentage of participants with Grade ≥ 3 Treatment-Emergent Adverse Events (TEAEs) that are treatment-related or Serious Adverse Events (SAEs) that are treatment-related in Part 1 and Part 2 of the study. | 16 Weeks
  The safety of VE202 and placebo in Parts 1 and 2 of the study, which include an 8-week and 2-week course of treatment, respectively, will be evaluated.

SECONDARY OUTCOMES:
Percentage of participants with endoscopic response on flexible sigmoidoscopy at Week 8, following treatment with VE202 for 2 weeks. | 8 Weeks
  Endoscopic response is defined as a reduction from baseline of 1 point or more in Mayo endoscopic subscore. The Mayo endoscopic subscore is evaluated on a scale of 0 to 3, with a higher score representing more severe disease.
Number of participants with TEAEs, SAEs, and Adverse Events of Special Interest (AESIs) in Parts 1, 2, and 3 of the study. | 52 Weeks
  The safety of VE202 and placebo in Parts 1, 2, and 3 of the study, which include an 8-week and 2-week course of treatment followed by a long-term follow-up period, will be evaluated. AESIs are defined as treatment-related Grade ≥2 TEAEs that are gastrointestinal or bacterial infections.
Percentage of participants with clinical remission at Week 8 of Part 1 and Week 8 of Part 2. | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. Clinical remission is defined as attaining a Mayo stool frequency subscore of ≤1 and an improvement in stool frequency subscore of ≥1 point from baseline, a rectal bleeding subscore of 0 and an endoscopic subscore ≤1. Each component of the Mayo score is evaluated on a scale of 0 to 3, with a higher score representing more severe disease.
Percentage of participants with clinical response at Week 8 of Part 1 and Week 8 of Part 2. | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. Clinical response is defined as having met the definition of clinical remission or having a decrease from baseline of ≥2 points and a decrease of ≥30% in modified Mayo score, with either a rectal bleeding score of 0 or a decrease in rectal bleeding of ≥1 point. Each component of the modified Mayo score (stool frequency, rectal bleeding, endoscopy findings) is evaluated on a scale of 0 to 3, with a higher score representing more severe disease.
Percentage of participants with endoscopic remission on flexible sigmoidoscopy at Week 8 of Part 1 and Week 8 of Part 2. | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. Endoscopic response is defined as a Mayo endoscopic subscore of 0 or 1 point. The Mayo endoscopic subscore is evaluated on a scale of 0 to 3, with a higher score representing more severe disease.
Change in Mayo score compared with baseline at Week 8 of Part 1 and Week 8 of Part 2. | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. The Mayo score is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician global assessment), with each parameter evaluated on a scale of 0 to 3. The total score ranges from 0 to 12, and a higher score represents more severe disease.
Histologic improvement at Week 8 of Part 1 and Week 8 of Part 2 as measured by Geboes score. | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. The Geboes score encompasses 6 dimensions, each with 4 subcategories: architectural changes, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in the epithelium, crypt destruction, and erosions or ulcerations. The Geboes score ranges from grade 0 to 5.4. A higher Geboes score represents more severe disease.
Histologic improvement at Week 8 of Part 1 and Week 8 of Part 2 as measured by the Robarts Histopathology Index (RHI). | 8 Weeks
  Participants will receive 8 weeks of VE202/placebo in Part 1 and 2 weeks of VE202/placebo in Part 2. The RHI provides a score between 0 and 33, based on the levels of chronic inflammatory infiltrate, neutrophils in lamina propria and epithelium, and erosion/ulceration. A higher RHI score represents more severe disease.
Change in fecal calprotectin levels after 2- and 8-week courses of VE202. | 52 Weeks
  The change in fecal calprotectin level from baseline will be evaluated.
Change in colonization with VE202 strains detected in feces at various time points in patients treated with 2- and 8-week courses of VE202. | 52 Weeks
  VE202 colonization will be characterized in patients treated with 2- and 8-week courses of VE202.
Change in the total percent of relative abundance of VE202 strains in feces at various time points in patients treated with 2- and 8-week courses of VE202. | 52 Weeks
  VE202 colonization will be characterized in patients treated with 2- and 8-week courses of VE202.
Change in taxonomic composition of gut microbiome in patients treated with 2- and 8-week courses of VE202. | 52 Weeks
  Microbiome composition will be evaluated by measuring the sum of species and the genera or higher-level taxonomic groupings at baseline and at subsequent time points in patients treated with 2- and 8-week courses of VE202 or placebo.
Change in fecal metabolite profiles at baseline and post-VE202 or placebo at various time points. | 52 Weeks
  Short-chain fatty acid and bile acid concentrations will be evaluated at baseline and at subsequent time points in patients treated with 2- and 8-week courses of VE202 or placebo.
Number of participants with hospitalization or surgical procedure related to UC after 2- and 8-week courses of VE202. | 52 weeks
  To evaluate the impact of 2- and 8-week courses of VE202 on Inflammatory bowel disease (IBD) specific healthcare resource utilization.
Change in patient-reported outcome measures using the Inflammatory Bowel Disease Questionnaire (IBDQ) to evaluate the impact of 2- and 8-week courses of VE202 IBD-specific health-related quality of life. | 52 Weeks
  The 32-item IBDQ uses a 7-point scale to assess disease-specific health-related quality of life across 4 dimensions: bowel symptoms, systemic symptoms, emotional wellbeing, and social function. The total IBDQ score is calculated by adding the scores within each domain. Scores can range from 32 to 224, with a higher score indicating a better outcome.
Change in patient-reported outcome measures using the EuroQoL-5D Health Assessment Questionnaire (EQ-5D) scores to evaluate the impact of 2- and 8-week courses of VE202 IBD-specific health-related quality of life. | 52 Weeks
  The EuroQoL-5D Health Assessment Questionnaire (EQ-5D) is a standardized, self-administered, non-disease-specific instrument for measuring generic health status for routine clinical outcome measurement in the delivery of operational healthcare. Scores range from 0 to 100, with a higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (10):
  - GI Pros Research, Naples, Florida
  - Revival Clinical Research, Orlando, Florida
  - Atlanta Center for Gastroenterology, P.C. & Atlanta Endoscopy Center, LTD, Decatur, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - NYU IBD Center, New York, New York
  - Cornell University Weill Cornell Medicine New York Presbyterian Hospital, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - Gastroenterology Research of America, LLC, San Antonio, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Misericordiae Ltd and Mater Research Ltd, South Brisbane, Queensland
  - St Vincent's Hospital Melbourne Department of Gastroenterology, Fitzroy, Victoria
- Bulgaria (2):
  - UMHAT Medica Ruse OOD, Rousse
  - Medical Centre Asklepion Main, Sofia
- Czechia (2):
  - Vojenská nemocnice Brno, Interní oddělení, Brno
  - PreventaMed s.r.o, Vila zdraví, Olomouc
- Hungary (3):
  - Semmelweis Egyetem Belgyógyászati és Hematológiai Klinika, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Dept. Gastroenterology, Univ. Debrecen, Debrecen
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Leiden University Medical Center, Leiden
- Poland (8):
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością Medic-R Spółka komandytowa, Poznan, Greater Poland Voivodeship
  - Medrise Sp. z o.o., Lublin, Lublin Voivodeship
  - MEDICAL NETWORK Sp. z o.o. WIP Warsaw IBD Point, Warsaw, Masovian Voivodeship
  - Centrum Medyczne "MEDYK", Rzeszów, Podkarpackie Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Vita Longa Sp. z o.o., Katowice
  - Solumed Centrum Medyczne, Poznan
  - Bonifraterskie Centrum Medyczne Sp. z o.o, Lodz, Łódź Voivodeship
- Ukraine (14):
  - M.Sklifosovsky Poltava Regional Clinical Hospital Regional Gastroenterology Center, Poltava, Poltavska
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Regional Clinical Hospital of the Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Municipal Nonprofit enterprise Kyiv City Clinical Hospital # 18, Kyiv
  - Artes Medikum, Medial Center, Llc, Kyiv
  - Medical Center OK!Clinic+, Kyiv
  - National Institute of Surgery and Transplantology named after O. O. Shalimova, Kyiv
  - LLC Medical Center "Consilium Medical", Kyiv
  - Volyn Regional Clinical hospital, Lutsk
  - Ternopil Regional Clinical Hospital, Ternopil
  - Uzhgorod City Multidisciplinary Clinical Hospital, Uzhhorod
  - Transcarpathian Regional Clinical Hospital named after Andria Novak, Uzhhorod
  - Vinnytsia Regional Clinical Hospital named after M.I. Pirogov, Vinnytsia
  - Vinnytsia City Clinical Hospital No. 1, Vinnytsia
- United Kingdom (4):
  - UHB NHSFT Queen Elizabeth Hospital, Birmingham, West Midlands
  - Barts Health NHS TrustThe Royal London Hospital, London
  - King's College Hospital, London
  - Imperial College Healthcare NHS Trust - St Mary's Hospital, London